CLINICAL TRIAL: NCT05760794
Title: BEST: Barbed-suture Efficiency Study for Sacrocolpopexy
Brief Title: Barbed-suture Efficiency Study for Sacrocolpopexy
Acronym: BEST
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00093867
Record Dates: First submitted 2023-02-25; First posted 2023-03-08 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Prolapse; Female
Keywords: sacrocolpopexy; pelvic organ prolapse; vaginal mesh attachment
MeSH Terms: conditions — Prolapse; Pelvic Organ Prolapse

STUDY DESIGN:
Intervention Model Description: Plan to enroll 52 participants with intention to treat 26 in each group - Participants will be randomized to delayed-absorbable barbed suture (2-0 V-Loc) versus delayed-absorbable interrupted suture (2-0 PDS).
Who Masked: Participant, Outcomes Assessor
Masking Description: Patient will be masked to their allocation and post-operative examiners will be masked at the 6 week, 6 month, and 12 month visits
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Non-barbed delayed absorbable suture (Experimental): Participants assigned to Non-barbed delayed absorbable suture group will have Non-barbed delayed absorbable suture used for vaginal mesh attachment at time of SCP
  Interventions: Procedure: Non-barbed delayed absorbable suture
- Barbed delayed absorbable suture (Experimental): Participants assigned to Barbed delayed absorbable suture group will have Barbed delayed absorbable suture used for vaginal mesh attachment at time of SCP
  Interventions: Procedure: Barbed delayed absorbable suture

INTERVENTIONS:
Procedure: Non-barbed delayed absorbable suture — The non-barbed delayed absorbable suture group vaginal mesh attachment will be performed with 2-0 PDS (polydioxanone). The vaginal mesh will be attached with at least four interrupted sutures on the anterior vagina and posterior vagina.
  Arms: Non-barbed delayed absorbable suture
Procedure: Barbed delayed absorbable suture — The barbed delayed absorbable suture group vaginal mesh attachment will be performed with 2-0 V-Loc. The vaginal mesh will be attached with a running V-Loc on the anterior and posterior vagina.
  Arms: Barbed delayed absorbable suture

SUMMARY:
Minimally invasive sacrocolpopexy (SCP) performed laparoscopically or with robotic assistance is associated with improved patient-centered outcomes such as faster recovery times, less pain, less bleeding, and shorter hospital stay, however at the expense of longer operating times. One of the time consuming parts of the procedure is vaginal mesh attachment.

DETAILED DESCRIPTION:
The purpose of this research study is to compare two different suture types that are used to attach vaginal mesh that is typically used in women undergoing robotic or laparoscopic sacrocolpopexy (attachment of the vagina to the sacral promontory). The barbed suture is one continuous suture, while the delayed absorbable suture involves placing individual sutures and tying a knot for each. All women will have permanent sutures that attach the mesh to the sacral promontory, which is standard of care. The goal is to determine if the barbed delayed absorbable suture decreases the time of vaginal mesh attachment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥21
* Subject must have apical with anterior or posterior vaginal prolapse with leading edge of prolapse to or beyond the hymen
* Subject reports a bothersome bulge they can see or feel per Pelvic Floor Disability Index (PFDI-20), question 3, response of 2 or higher
* Eligible for laparoscopic or robotic sacrocolpopexy
* Desires surgical treatment for symptomatic uterovaginal or vaginal vault prolapse
* English speaking

Exclusion Criteria:

* Patients who are not surgical candidates due to medical comorbidities
* Current foreign body complications (including but not limited to erosion, fistula, abscess). This covers foreign bodies of any type (e.g. synthetic and biologic including allograft, xenograft).
* Inability to give informed consent or to complete the testing or data collection.
* Anticipated circumstances resulting in an inability to follow up (geographic relocation, etc.).
* Active systemic infection including any gynecologic infection, untreated Urinary Tract Infection (UTI) or tissue necrosis.
* History of pelvic organ cancer (e.g. uterine, ovarian, bladder, or cervical).
* Prior or currently undergoing radiation, laser therapy, or chemotherapy in the pelvic area.
* Subject has taken systemic steroids (within the last month, steroid inhalers OK), or immunosuppressive or immunomodulatory treatment (within the last 3 months)
* Systemic connective tissue disease (e.g. scleroderma, Marfan's syndrome, Ehlers Danhlos, collagenosis, polymyositis or polymyalgia rheumatic, lupus)
* Chronic systemic pain that includes the pelvic area or chronic focal pain that involves the pelvis
* Poorly controlled diabetes mellitus (DM), as indicated by Hemoglobin A1c > 9
* Those requiring concomitant rectopexy
* Subject is not able to conform to steep Trendelenburg position
* Known sensitivity to polypropylene
* History of prior prolapse repair utilizing vaginal or abdominal mesh
* Planned vaginal mesh attachment placed transvaginally
* History of diverticulitis

Ages: 21 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — women with symptomatic uterovaginal or vaginal vault prolapse, without a prior history of mesh repair, who have completed childbearing, are seeking surgical management, and are willing to proceed with abdominal placement of permanent synthetic mesh.
Enrollment: 52 (Estimated)
Dates: Start 2023-06-21 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Time to complete vaginal graft attachment | Day 1
  To determine if delayed-absorbable barbed suture (2-0 V-Loc) produces a decrease in the time to achieve vaginal mesh attachment during minimally invasive SCP (with or without concomitant total hysterectomy) compared to delayed- absorbable polydioxanone (2-0 PDS) interrupted suture - time (in minutes and seconds)

SECONDARY OUTCOMES:
Composite success rate | Year 1
  To compare the 1-year composite success rates of minimally invasive sacrocolpopexy (SCP) between the two groups:
  * Anatomic success: leading edge of prolapse is at or above the hymen (POP-Q point Ba and Bp less than or equal to and vaginal apex less than 1/3 of the total vaginal length
  * Subjective success: patient denies symptoms of vaginal bulging per Pelvic Floor Distress Inventory (PFDI)-20 question 3, answering "No" or "Yes" but "Not at all" bothersome
  * Assessment for re-intervention or re-operation for recurrence or persistence of pelvic organ prolapse: No need for pessary use or additional surgical treatment for prolapse at any time after the initial procedure
Vaginal mesh exposure at 1 year | Year 1
  To compare the 1 year rate of vaginal mesh exposure between the two groups - Signs and symptoms of mesh exposure include vaginal or pelvic pain, vaginal discharge or bleeding, odor, recurrent infection, abscess development, dyspareunia, or pain experienced by the sexual partner. Pain is the most common presenting symptom.
Adverse outcome scores | Week 6
  To compare adverse outcomes, classified according to the Clavien-Dindo system, between the two groups - It consists of 7 grades (I, II, IIIa, IIIb, IVa, IVb and V) - the higher the grade; the worse the complication
Surgeon satisfaction with technique | Day 1
  To compare intraoperative surgeon satisfaction with technique between the two groups - satisfaction with technique will be assessed with a 10 point visual analog scale (VAS) for ease of placement, appearance of mesh attachment, and global satisfaction with the attachment type - 0 meaning difficult and 10 meaning easy
Patient change in quality of life, symptom bother, and sexual functioning - (PFDI-20) Pelvic Floor Distress Inventory | Year 1
  Assessment of participant changes in quality of life, symptom bother, and sexual functioning at 1 year compared to baseline - The total PFDI-20 score was classified as the absence of symptoms (score zero), symptoms with mild distress (1 to 15 points), symptoms with moderate distress (16 to 34 points), and symptoms with severe distress (35 to 40 points)
Patient change in quality of life, symptom bother, and sexual functioning - (PISQ-sf) Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire short form | Year 1
  Assessment of participant changes in quality of life, symptom bother, and sexual functioning at 1 year compared to baseline - a validated general questionnaire widely used in clinical practice as a screening tool for female sexual dysfunction, as well as in clinical trials as an outcome measure. It consists of 19 items, grouped into six domains: Desire, Arousal, Lubrication, Orgasm, Satisfaction, and Pain. The total score is obtained by adding the six domain scores (range: 2.0-36.0). Higher scores in particular domains and total score indicate better sexual function.
Patient change in quality of life, symptom bother, and sexual functioning - (PFIQ-sf7) Pelvic Floor Impact Questionnaire Short form | Year 1
  Assessment of participant changes in quality of life, symptom bother, and sexual functioning at 1 year compared to baseline - scores range from 0-300. A lower score means there is a lesser effect on quality of life.

OTHER OUTCOMES:
Mesh related adverse events and surgical success compared to PACT trial | Year 1
  To compare mesh-related adverse events (mesh exposure, pain) and surgical success within the first post-operative year in the BEST trial compared to historical data collected in the PACT trial.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine L Woodburn, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maher C, Feiner B, Baessler K, Schmid C. Surgical management of pelvic organ prolapse in women. Cochrane Database Syst Rev. 2013 Apr 30;(4):CD004014. doi: 10.1002/14651858.CD004014.pub5. PMID 23633316
- [Background] Siddiqui NY, Grimes CL, Casiano ER, Abed HT, Jeppson PC, Olivera CK, Sanses TV, Steinberg AC, South MM, Balk EM, Sung VW; Society of Gynecologic Surgeons Systematic Review Group. Mesh sacrocolpopexy compared with native tissue vaginal repair: a systematic review and meta-analysis. Obstet Gynecol. 2015 Jan;125(1):44-55. doi: 10.1097/AOG.0000000000000570. PMID 25560102
- [Background] Paraiso MF, Walters MD, Rackley RR, Melek S, Hugney C. Laparoscopic and abdominal sacral colpopexies: a comparative cohort study. Am J Obstet Gynecol. 2005 May;192(5):1752-8. doi: 10.1016/j.ajog.2004.11.051. PMID 15902189
- [Background] Geller EJ, Siddiqui NY, Wu JM, Visco AG. Short-term outcomes of robotic sacrocolpopexy compared with abdominal sacrocolpopexy. Obstet Gynecol. 2008 Dec;112(6):1201-1206. doi: 10.1097/AOG.0b013e31818ce394. PMID 19037026
- [Background] Matthews CA, Geller EJ, Henley BR, Kenton K, Myers EM, Dieter AA, Parnell B, Lewicky-Gaupp C, Mueller MG, Wu JM. Permanent Compared With Absorbable Suture for Vaginal Mesh Fixation During Total Hysterectomy and Sacrocolpopexy: A Randomized Controlled Trial. Obstet Gynecol. 2020 Aug;136(2):355-364. doi: 10.1097/AOG.0000000000003884. PMID 32649494
- [Background] Bazzi AA, Osmundsen BC, Hagglund KH, Aslam MF. Anatomical Outcomes Based on Suturing Technique During Vaginal Mesh Attachment in Robotic Sacrocolpopexy. Female Pelvic Med Reconstr Surg. 2019 Mar/Apr;25(2):105-108. doi: 10.1097/SPV.0000000000000654. PMID 30807409
- [Background] Moore R, Moriarty C, Chinthakanan O, Miklos J. Laparoscopic sacrocolpopexy: operative times and efficiency in a high-volume female pelvic medicine and laparoscopic surgery practice. Int Urogynecol J. 2017 Jun;28(6):887-892. doi: 10.1007/s00192-016-3179-1. Epub 2016 Oct 20. PMID 27766346
- [Background] Catanzarite T, Saha S, Pilecki MA, Kim JY, Milad MP. Longer Operative Time During Benign Laparoscopic and Robotic Hysterectomy Is Associated With Increased 30-Day Perioperative Complications. J Minim Invasive Gynecol. 2015 Sep-Oct;22(6):1049-58. doi: 10.1016/j.jmig.2015.05.022. Epub 2015 Jun 10. PMID 26070725
- [Background] Childers CP, Maggard-Gibbons M. Understanding Costs of Care in the Operating Room. JAMA Surg. 2018 Apr 18;153(4):e176233. doi: 10.1001/jamasurg.2017.6233. Epub 2018 Apr 18. PMID 29490366
- [Background] Crane AK, Geller EJ, Matthews CA. Trainee performance at robotic console and benchmark operative times. Int Urogynecol J. 2013 Nov;24(11):1893-7. doi: 10.1007/s00192-013-2102-2. Epub 2013 May 3. PMID 23640003
- [Background] Tan-Kim J, Nager CW, Grimes CL, Luber KM, Lukacz ES, Brown HW, Ferrante KL, Dyer KY, Kirby AC, Menefee SA. A randomized trial of vaginal mesh attachment techniques for minimally invasive sacrocolpopexy. Int Urogynecol J. 2015 May;26(5):649-56. doi: 10.1007/s00192-014-2566-8. Epub 2014 Nov 25. PMID 25421934
- [Background] Lowman JK, Woodman PJ, Nosti PA, Bump RC, Terry CL, Hale DS. Tobacco use is a risk factor for mesh erosion after abdominal sacral colpoperineopexy. Am J Obstet Gynecol. 2008 May;198(5):561.e1-4. doi: 10.1016/j.ajog.2008.01.048. Epub 2008 Apr 2. PMID 18377864
- [Background] Cundiff GW, Varner E, Visco AG, Zyczynski HM, Nager CW, Norton PA, Schaffer J, Brown MB, Brubaker L; Pelvic Floor Disorders Network. Risk factors for mesh/suture erosion following sacral colpopexy. Am J Obstet Gynecol. 2008 Dec;199(6):688.e1-5. doi: 10.1016/j.ajog.2008.07.029. Epub 2008 Oct 31. PMID 18976976
- [Background] Tan-Kim J, Menefee SA, Luber KM, Nager CW, Lukacz ES. Prevalence and risk factors for mesh erosion after laparoscopic-assisted sacrocolpopexy. Int Urogynecol J. 2011 Feb;22(2):205-12. doi: 10.1007/s00192-010-1265-3. Epub 2010 Sep 15. PMID 20842494
- [Derived] Gabra M, Woodburn KL, El Haraki A, Zdroik A, Duong M, Mezes C, Fisher M, Paukner L, Matthews CA. BEST: Barbed-suture Efficiency Study for Sacrocolpopexy: A Randomized Clinical Trial. Urogynecology (Phila). 2025 Nov 12. doi: 10.1097/SPV.0000000000001768. Online ahead of print. PMID 41252163